CLINICAL TRIAL: NCT02839876
Title: Comparison of Multimodal Analgesic Regimen With Intravenous Acetaminophen to Standard Oral Multimodal Therapy in Primary Total Hip Arthroplasty: A Randomized Controlled Double Blind Trial
Brief Title: Intravenous Versus Oral Acetaminophen in Primary Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00072610
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis; Acetaminophen; Arthroplasty, Hip Replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous acetaminophen (Experimental): Subjects receive 1000 mg acetaminophen IV immediately preoperatively, as well as at 6, 12, and 18 hours postoperatively. At the same time points, subjects will receive an oral placebo.
  Interventions: Drug: Intravenous acetaminophen
- Oral acetaminophen (Active Comparator): Subjects receive 1000 mg acetaminophen PO immediately preoperatively, as well as at 6, 12, and 18 hours postoperatively. At the same time points, subjects will receive an intravenous placebo.
  Interventions: Drug: Oral acetaminophen

INTERVENTIONS:
Drug: Intravenous acetaminophen — Subject receives 1 g acetaminophen by the intravenous route every 6 hours for 4 doses beginning in the preoperative holding area.
  Other Names: Ofirmev
  Arms: Intravenous acetaminophen
Drug: Oral acetaminophen — Subject receives 1 g acetaminophen by the oral route every 6 hours for 4 doses beginning in the preoperative holding area.
  Arms: Oral acetaminophen

SUMMARY:
The purpose of this study is to determine if intravenous acetaminophen is superior to oral acetaminophen when used as part of a multimodal pathway for primary total hip arthroplasty.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized controlled study. 60 subjects will be recruited (see #6 Recruitment and Compensation below). On the day of surgery, subjects will be randomized to receive either the study intervention (intravenous acetaminophen and placebo tablets) or the control intervention (intravenous saline and active acetaminophen tablets). The Investigational Drug Service will prepare each intervention package, which will include one intravenous and one oral medication dose. Only one of these routes will be active (determined by randomization). Subjects will receive doses of both an intravenous and oral study drug every 6 hours in order to maintain blinding, and will receive a total of 4 doses of each (at 0, 6, 12 and 18 hours). The dose of acetaminophen in all cases will be 1000 mg. The volume of intravenous acetaminophen (and saline) will be 100 mL. The oral dose will consist of two (2) tablets of 500 mg each (or two matching placebo tablets).

All subjects will receive a standardized anesthetic regimen for total hip arthroplasty, as follows:

A) Preoperative phase

Subjects will receive the following preoperative multimodal drugs:

* Pregabalin 75 mg PO
* Celecoxib 200 mg PO
* The interventional drugs, both IV and PO . The time that these drugs are administered will be recorded as time zero. Patients will then receive a spinal anesthetic with 12.5 mg of isobaric bupivacaine. No peripheral nerve blocks will be performed.

B) Intraoperative phase All subjects will be receive propofol infusion beginning at 50 mg/kg/min and titrated to a Richmond Agitation-Sedation Scale score of -1 to -3 (drowsy to moderate sedation). Dexamethasone 10 mg IV and ketamine 0.25 mg/kg IV up to 40 mg total will be administered as part of the standard multimodal regimen. If required, subjects may receive fentanyl 25 mcg IV as needed to treat discomfort. No joint infiltration will be performed by the surgeon.

C) Postoperative phase In the Post-Anesthesia Care Unit (PACU), subjects will have an intravenous patient-controlled analgesia (IVPCA) device connected and loading doses of hydromorphone administered by the PACU nurse as necessary (0.2 mg q 8 min prn).

On the floor, subjects will receive:

* Pregabalin 75 mg PO BID until discharge
* Celecoxib 200 mg PO BID until discharge
* Dexamethasone 10 mg IV x 1 on postoperative day 1 (24 hours after the first dose)
* Intravenous patient-controlled analgesia (IVPCA) with hydromorphone (0.2 mg q 8 min).

The remaining 3 intervention packages (IV and PO) will be administered at 6, 12 and 18 hours following the first dose. At time point 24 hours (i.e. the fifth dose of acetaminophen), all subjects will begin to receive 975 mg of oral acetaminophen, continuing every six hours until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective, primary total hip replacement for osteoarthritis
* American Society of Anesthesiologists (ASA) Physical Classification I-III
* Weight 50 kg or greater
* Body mass index 18-40 kg/m2

Exclusion Criteria:

* Inability to consent to study
* Inability to speak English
* Pregnancy
* Weight <50 kg
* Revision hip replacement or emergency surgery
* Contraindications to spinal anesthesia: coagulopathy or bleeding diathesis, local infection, allergy to local anesthetics
* Allergies/intolerances/contraindications to any of the multimodal agents: acetaminophen, pregabalin, celecoxib, ketamine, or dexamethasone
* Chronic pain from a separate source other than operative hip
* Daily opioid equivalent use of 30 mg of morphine or greater at time of consent
* History of heart failure
* History of drug or alcohol abuse
* Rheumatoid arthritis
* Uncontrolled anxiety, schizophrenia or other psychiatric disorder that, in the opinion of the investigator, may interfere with the study assessments
* Chronic malnutrition, renal or liver impairment
* Hypersensitivity to acetaminophen or any of its excipients

Ages: 56 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Started | 41 | 40
Completed | 31 | 29
Not Completed | 10 | 11
Not completed — Protocol Violation | 10 | 11

BASELINE CHARACTERISTICS:
Population: Only completed participants are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 65 [61 to 71] | 63 [59 to 67] | 64.5 [60.5 to 70.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 21 | 13 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 23 | 23 | 46
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
ASA Physical Classification [Count of Participants; unit: Participants] — Participants were classified per the American Society of Anesthesiologists (ASA) Physical Class I-III. ASA I = A normal healthy patient; ASA II = A patient with mild systemic disease; ASA III = A patient with severe systemic disease
  Participants
    ASA I | 1 | 0 | 1
    ASA II | 17 | 19 | 36
    ASA III | 13 | 10 | 23
Weight [Mean (Standard Deviation); unit: kilograms] | 87.99 (21.90) | 87.25 (18.79) | 87.63 (20.29)

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Opioid Consumption
Description: Cumulative dose of hydromorphone consumed in the first 24 hours postoperatively
Time Frame: 24 hours
Population: Only completed participants are included.
Measure: Median (Inter-Quartile Range); unit: morphine milliequivalent
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
morphine milliequivalent | 3.0 [1.9 to 6.0] | 3.4 [2.0 to 5.9]

2. Secondary Outcome: Opioid Consumption (Other)
Description: morphine equivalent units of intravenous and oral opioids
Time Frame: 0-48 hours
Measure: Median (Inter-Quartile Range); unit: morphine milliequivalent
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
morphine milliequivalent | 6.2 [3.0 to 12.1] | 6.8 [3.9 to 11.7]

3. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (Preoperatively)
Description: Pain scores (using NRS-11 scale) with active range of motion of the hip. Participants rate their pain on an 11-point scale (0=no pain at all, 10=worst imaginable pain).
Time Frame: preoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 7.0 [5.0 to 8.0] | 7.0 [6.0 to 8.0]

4. Secondary Outcome: Pain Scores, as Measured by the 11-point Numeric Rating Scale (NRS-11) (1 Hour After Arrival to PACU)
Description: Pain scores (using NRS-11 scale) at rest. Participants rate their pain on an 11-point scale (0=no pain at all, 10=worst imaginable pain).
Time Frame: 1 hour after arrival to PACU
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 1.0 [0.0 to 3.75] | 1.0 [0.0 to 3.0]

5. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (8 Hours)
Description: as for outcome 4
Time Frame: 8 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 2.0 [0.0 to 4.75] | 3.0 [0.0 to 5.0]

6. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (24 Hours)
Description: as for outcome 4
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 2.0 [1.0 to 3.5] | 1.0 [0.0 to 3.0]

7. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (36 Hours)
Description: as for outcome 4
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 3.0 [1.0 to 4.0] | 2.0 [0.75 to 3.0]

8. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (48 Hours)
Description: as for outcome 4
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 2.0 [1.0 to 3.0] | 2.0 [0.0 to 3.0]

9. Secondary Outcome: Subject Satisfaction at 24 Hours
Description: Overall subject satisfaction with hospital experience at the 24 hour time point using a simple 11-point Likert scale to quantify global satisfaction. 0=completely unsatisfied, 10=completely satisfied.
Time Frame: 24 hours
Population: Only completed participants are included.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 9 [8 to 10] | 9 [8 to 10]

10. Secondary Outcome: Subject Satisfaction at 48 Hours (48 Hours)
Description: Overall subject satisfaction with hospital experience at the 48 hour time point using a simple 11-point Likert scale to quantify global satisfaction. 0=completely unsatisfied, 10=completely satisfied.
Time Frame: 48 hours
Population: Only completed participants are included.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 9 [8 to 10] | 9 [9 to 10]

11. Secondary Outcome: Straight Leg Raise
Description: Number of participants who are able to complete the active straight leg test. The subject rests supine and is asked to lift his/her operative lower limb (with knee extended) until the ankle is 20 cm from level. If the subject can do this, the test is positive.
Time Frame: Postoperative day 1
Population: Only completed participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
Participants | 16 | 11

12. Secondary Outcome: Heel Slide Test
Description: Number of participants who are able to complete the heel-slide test. The subject rests supine and is asked to place the heel of his/her operative side on the contralateral knee, then slide the heel down to the ankle and back in one continuous motion. If the subject can do this, the test is positive. If the subject cannot do this in one motion, or if pain or other factors prevent the test from being performed, the test is negative.
Time Frame: Postoperative day 1
Population: Only completed participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
Participants | 25 | 16

13. Secondary Outcome: Number of Participants Able to Complete the Supine to Sit Test
Description: Number of participants able to go from supine to a sitting position independently.
Time Frame: Postoperative day 1
Population: Only completed participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
Participants | 10 | 6

14. Secondary Outcome: Self-paced Walk Test
Description: Time taken to walk down a hallway 20 m at a safe and quick pace, turn around and return to starting point.
Time Frame: Postoperative day 1
Population: Only completed participants are included.
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
seconds | 86 [41 to 1641] | 63 [43 to 1328]

15. Secondary Outcome: Number of Participants With Opioid-related Adverse Events
Description: Incidence of respiratory desaturation events, nausea, vomiting, pruritis, ileus, and constipation
Time Frame: 0-72 hours
Population: Only completed participants are included.
Measure: Number; unit: participants
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
participants | 15 | 7

16. Secondary Outcome: Analgesic Consumption as Measured by Patient Diary
Description: morphine equivalent units of oral opioids and other non-opioids
Time Frame: day 30
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
mg | 0 [0 to 0] | 0 [0 to 0]

17. Secondary Outcome: Worst Pain (Day 30)
Description: Participants are asked to rate their WORST pain on POSTOPERATIVE DAY 30 on an 11-point scale (0=no pain at all, 10=worst imaginable pain).
Time Frame: day 30
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 1.0 [0.0 to 2] | 0 [0 to 3]

18. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (Preoperatively)
Description: as for outcome 4
Time Frame: preoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 1.0 [0.0 to 4.0] | 2.0 [0.0 to 5.0]

19. Secondary Outcome: Pain Scores, as Measured by the 11-point Numeric Rating Scale (NRS-11) (1 Hour After Arrival to PACU)
Description: Pain scores (using NRS-11 scale) at with active range of motion of the hip. Participants rate their pain on an 11-point scale (0=no pain at all, 10=worst imaginable pain).
Time Frame: 1 hour after arrival to PACU
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 2.0 [0.0 to 4.75] | 2.0 [0.0 to 4.0]

20. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (8 Hours)
Description: as for outcome 3
Time Frame: 8 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 3.0 [1.0 to 5.0] | 5.5 [3.75 to 7.25]

21. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (24 Hours)
Description: as for outcome 3
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 5.0 [3.0 to 7.5] | 4.0 [3.0 to 7.0]

22. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (36 Hours)
Description: as for outcome 3
Time Frame: 36 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 5.0 [3.0 to 70] | 4.5 [3.75 to 6.0]

23. Secondary Outcome: Subject Satisfaction at 48 Hours
Description: as for outcome 10
Time Frame: 48 hours
Population: Only completed participants are included.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 9 [8 to 10] | 9 [9 to 10]

24. Secondary Outcome: Pain Score, as Measured by the 11-point Numeric Rating Scale (NRS-11) (48 Hours)
Description: as for outcome 3
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
score on a scale | 5.0 [3.0 to 6.0] | 5.0 [2.5 to 6.0]

25. Other Pre Specified Outcome: Hospital Length of Stay
Description: Time to both discharge readiness and to actual discharge
Time Frame: 0-72 hours
Population: Only completed participants are included.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
days | 1 [1 to 2] | 1 [1 to 2]

26. Other Pre Specified Outcome: Overall Hospital Admission Costs
Description: difference in total hospital admission cost between groups
Time Frame: 0-72 hours
Measure: Median (Inter-Quartile Range); unit: US dollars
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
US dollars | 14682 [13468 to 16353] | 14782 [13461 to 17013]

27. Other Pre Specified Outcome: Pharmacy-related Costs
Description: difference in pharmacy-related cost between groups
Time Frame: 0-72 hours
Measure: Median (Inter-Quartile Range); unit: US dollars
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
US dollars | 498 [465 to 518] | 510 [459 to 539]

28. Other Pre Specified Outcome: Costs Related to Opioid-related Adverse Events
Description: difference in cost related to treatment of opioid-related adverse events (nausea, vomiting, pruritis, constipation, respiratory depression, dizziness) between groups
Time Frame: 0-72 hours
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
US dollars | 0.80 (1.18) | 0.85 (1.73)

29. Other Pre Specified Outcome: Cost Associated With Nursing Interventions and Drugs to Treat Opioid-related Adverse Events
Description: mean cost (per patient) related to nursing care of opioid-related adverse events (nausea, vomiting, pruritis, constipation, respiratory depression, dizziness) in $USD
Time Frame: 0-72 hours
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
Number analyzed (Participants) | 31 | 29
US dollars | 1.86 (2.68) | 1.82 (3.50)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Intravenous Acetaminophen | Oral Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/29
Other Adverse Events (participants affected / at risk) | 13/31 | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Acetaminophen (N=31) | Oral Acetaminophen (N=29)
Postoperative hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — Postoperative infected hematoma, admitted to hospital, treated with surgery and antibiotics
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Acetaminophen (N=31) | Oral Acetaminophen (N=29)
Nausea (Gastrointestinal disorders) | 9 (10) | 3 (3)
constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
wound erythema/drainage (Infections and infestations) | 1 (1) | 3 (3)
Dizziness/orthostasis (Cardiac disorders) | 7 (7) | 1 (1)
Hip dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abnormal lab values (INR) (Investigations) | 1 (1) | 0 (0)
Polyneuropathy, peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT02839876/Prot_SAP_000.pdf